CLINICAL TRIAL: NCT00384098
Title: A Randomized, Double-blind, Parallel-group, 4-arm, 12-week Study to Evaluate the Safety and Efficacy of Topically Applied CTA018 vs Vehicle for the Treatment of Adult Subjects With Chronic Plaque Psoriasis
Brief Title: Safety and Efficacy of Topically Applied CTA018 in Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTA018-CL-2001
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2007-06

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CTA018 cream

SUMMARY:
Vitamin D and its analogs are currently widely used for the treatment of psoriasis. The study drug (CTA018) is a novel analog of vitamin D, and this Phase 2 study will investigate the efficacy and safety of CTA018 in the treatment of psoriasis. Patients with chronic plaque psoriasis will receive one of three doses of CTA018 cream or vehicle (no study drug) daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic plaque psoriasis for 6 months to a max 15% body surface area excluding face, scalp, groin, axillae, palms, soles of feet
* at least two evaluable plaques with CPSS >/= 6
* baseline PSGA >/= 2
* women of childbearing potential msut agree to use an effective form of contraception

Exclusion Criteria:

* cannot have guttate, pustular, erythrodermic or other non-plaque forms of psoriasis
* cannot have concomitant serious illness/condition that may interfere with participation in the study
* cannot have used topical therapy within 2 weeks prior to baseline visit
* cannot have used photo-therapy or systemic psoriasis therapy within 4 weeks prior to baseline visit
* cannot have had prolonged exposure to natural or artificial UV radiation within 4 weeks of baseline visit or intend to have exposure during the study
* cannot have used systemic immunomodulatory therapy within 12 weeks prior to baseline visit
* cannot have a history of hypercalcemia or kidney stones
* cannot be unable or unwilling to discontinue calcium and/or vitamin D supplementation during the study
* cannot be pregnant or a nursing mother
* cannot be participating in or have participated in an interventional study within 30 days of study start

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be treatment success or failure based on a Physician's Static Global Assessment (PSGA) of 0 or 1 (success).

SECONDARY OUTCOMES:
Secondary efficacy outcomes include time to success (PSGA), change in overall PSGA score, and Area Adjusted Psoriasis Area and Severity Index (AAPASI)changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Melnick, MD, Study Director — OPKO Renal
Locations (16):
- United States (16):
  - Radiant Research, Tucson, Arizona
  - Dermatology Research of Arkansas PLLC, Little Rock, Arkansas
  - Northwestern University, Chicago, Illinois
  - Radiant Research, Kansas City, Overland Park, Kansas
  - Mass General/ Brigham & Women's, Boston, Massachusetts
  - Department of Dermatology, Mayo Clinic, Rochester, Minnesota
  - UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Buffalo Medical Group PC, Williamsville, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Paddington Testing Co., Philadelphia, Pennsylvania
  - Radiant Research Inc., Anderson, South Carolina
  - Palmetto Clinical Trial Services LLC, Greenville, South Carolina